CLINICAL TRIAL: NCT05653271
Title: A Phase 1 Multicenter Study Evaluating the Safety and Efficacy of ACE1831, an Allogeneic Anti-CD20 Antibody-Conjugated Gamma Delta T-cell Therapy, in Adult Subjects With Relapsed/Refractory CD20-expressing B-cell Malignancies
Brief Title: ACE1831 in Adult Subjects With Relapsed/ Refractory CD20-expressing B-cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Acepodia Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACE1831-001
Record Dates: First submitted 2022-11-02; First posted 2022-12-16 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: B-cell Lymphoma; Non Hodgkin Lymphoma; DLBCL; Primary Mediastinal Large B Cell Lymphoma; Marginal Zone Lymphoma; Follicular Lymphoma; Burkitt Lymphoma; High-grade B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Burkitt Lymphoma | interventions — Cyclophosphamide; fludarabine; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group A (ACE1831) (Experimental): ACE1831 dose escalation, monotherapy. Lymphodepleting regimen followed by escalating doses of ACE1831.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: ACE1831
- Treatment Group B (ACE1831 and obinutuzumab) (Experimental): ACE1831 dose escalation, in combination with obinutuzumab. Lymphodepleting regimen followed by escalating doses of ACE1831, given in combination with obinutuzumab.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: ACE1831; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Cyclophosphamide — Lymphodepleting agent
Drug: Fludarabine — Lymphodepleting agent
Drug: ACE1831 — Allogeneic gamma delta T (gdT) cell therapy
Drug: Obinutuzumab — Anti-CD20 monoclonal antibody
  Arms: Treatment Group B (ACE1831 and obinutuzumab)

SUMMARY:
ACE1831 is an off-the-shelf, allogeneic gamma delta T (gdT) cell therapy derived from healthy donors, that is under investigation for the treatment of CD20-expressing B-cell malignancies.

The ACE1831-001 study is an open-label, Phase I, first-in-human (FIH) study that aims to evaluate the safety and tolerability, pharmacokinetics and pharmacodynamics, and efficacy of ACE1831 in patients with CD20-expressing Non-Hodgkin lymphoma.

ELIGIBILITY:
Key Inclusion Criteria:

* CD20-positive B-cell NHL that is persistent or progressive after having received at least 2 prior systemic therapies per NCCN guidelines
* At least 1 measurable lesion according to the revised International Working Group (IWG) Response Criteria for Malignant Lymphoma
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 or subjects with ECOG scores of 2 with a serum albumin of >3.5
* Adequate hematologic and renal, hepatic, and cardiac function
* Oxygen saturation via pulse oxygenation ≥ 92% at rest on room air

Key Exclusion Criteria:

* Prior treatment with a genetically modified cell therapy product targeting CD20
* Autologous stem cell transplant within 6 weeks of informed consent or history of allogeneic stem cell transplantation
* History of central nervous system (CNS) lymphoma or primary CNS lymphoma
* History or presence of clinically relevant CNS disorder (e.g. epilepsy)
* Clinically significant active infection
* Currently active, clinically significant cardiovascular disease
* Human Immunodeficiency virus (HIV) infection (however, subjects on anti-retroviral therapy for at least 4 weeks and with HIV viral loads of <400 copies/mL are eligible), active hepatitis B infection, or hepatitis C infection
* History of other malignancies with the exception of certain treated malignancies with no evidence of disease
* Primary immunodeficiency disorder
* Pregnant or lactating female
* Any medical, psychological, familial, or sociological conditions that, in the opinion of the Investigator or Sponsor Medical Monitor, would impair the ability of the subject to receive study treatment, comply with study requirements, or understanding of the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-01-21 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs), Dose Limiting Toxicities (DLTs), adverse events of special interest (AESIs), and serious adverse events (SAEs) | 2 years
Change from baseline in ECOG status | 1 year
Change from baseline in physical examination results | 1 year
  Number of subject with change from baseline clinically significant physical examination findings by dose level (descriptive)
Change from baseline clinical laboratory tests results | 1 year
  Number of subjects with change from baseline clinically significant lab findings by dose level (descriptive)
Change from baseline in urinalysis results | 1 year
  Number of subjects with change from baseline clinically significant urinalysis findings by dose level (descriptive)
Change from baseline in vital signs results | 1 year
  Number of subjects with change from baseline clinical significant vital signs findings by dose level (descriptive)
Change from baseline in electrocardiogram (ECG) results | 1 month
  Number of subjects with change from baseline clinically significant ECG findings by dose level (descriptive)
Maximum Tolerated Dose (MTD) | 1 month

SECONDARY OUTCOMES:
Persistence of ACE1831 after administration | 1 month
  Half-life of ACE1831
Measure of anti-ACE1831 antibodies after administration | 1 month
  Titration of anti-ACE1831 antibodies after administration
Objective Response Rate (ORR) | 2 years
  Objective response of each patient's underlying lymphoma, duration of response, and progression-free survival all based on the revised IWG Response Criteria for Malignant Lymphoma

OTHER OUTCOMES:
Pharmacodynamics of ACE1831 | 2 years
  Serum levels of interferon-γ, TNF-α, IL-2, IL-6, IL-8 and IL-10, as well as other potential biomarkers

CONTACTS AND LOCATIONS:
Locations (13):
- United States (5):
  - AdventHealth Orlando, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Queen Mary Hospital, Hong Kong, Hong Kong
- Taiwan (7):
  - Kaohsiung Chang-Gung Memorial Hospital, Kaohsiung City
  - Ministry of Health and Welfare Shuang-Ho Hospital, New Taipei City
  - Tamsui MacKay Memorial Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Linkou Chang-Gung Memorial Hospital, Taoyuan

IPD SHARING:
Plan to Share IPD: No